CLINICAL TRIAL: NCT02312752
Title: Intra-epidermal Stimulation (IES) of Small Nerve Fibers (A-delta Fibers)
Acronym: IES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Electrodes required gas sterilization before re-use which was not feasible
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 140103
Record Dates: First submitted 2014-11-12; First posted 2014-12-09 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Intra-epidermal stimulation in healthy control subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-epidermal stimulation (Other): A small piece of plastic with a tiny sharp protruding tip (the intra-epidermal stimulation electrode) will be applied to the foot and hand. Small "sticker" electrodes will be placed over nerves on the forearm or ankle. A stimulus will be applied to the electrode for intra-epidermal stimulation. The stimulus will be gradually increased from no stimulus to a stimulus that is barely felt as a pin-prick type of sensation. Thereafter, the stimulus will be applied 5-15 times per second for 10 periods of 40-60 seconds.
  Interventions: Device: Intra-epidermal stimulation electrode

INTERVENTIONS:
Device: Intra-epidermal stimulation electrode — A small piece of plastic with a tiny sharp protruding tip (the intra-epidermal stimulation electrode) will be applied to the foot and hand. Small "sticker" electrodes will be placed over nerves on the forearm or ankle. A stimulus will be applied to the electrode for intra-epidermal stimulation. The stimulus will be gradually increased from no stimulus to a stimulus that is barely felt as a pin-prick type of sensation. Thereafter, the stimulus will be applied 5-15 times per second for 10 periods of 40-60 seconds.

SUMMARY:
The purpose of the study is to determine whether a particular type of nerve fibers, A-delta fibers, can be tested in an Electromyography (EMG) lab on a routine basis. Normal, healthy volunteers will be enrolled in this study.

DETAILED DESCRIPTION:
The epidermis is the outermost layer of the skin that includes skin cells and small nerve fibers called A-delta fibers. A-delta fibers send signals to the brain about pin-prick type of pain and temperature. The investigators want to study whether the investigators can stimulate A-delta fibers and document this by recording electrical potentials from the nerves in subjects' limbs.

Study Procedures:

A small piece of plastic will be applied to your foot and your hand. A tiny sharp tip protrudes from this piece of plastic. You will be barely able to feel this sharp tip when touching the piece of plastic. This is the electrode for intra-epidermal stimulation.

With stimulation, you will feel a pin-prick type of sensation. The stimulus will be adjusted so that you barely feel the pin-prick type of sensation. The investigators will record responses of stimulation from nerves in your skin.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 21 through 60 years with no history or clinical signs of neuropathy.

Exclusion Criteria:

1. History of peripheral nerve disease or disease of somatosensory pathways.
2. Abnormalities on neurologic examination.
3. Prior or current exposure to known neurotoxins, such as excessive alcohol use or chemotherapy.
4. Neurologic or psychiatric conditions that would prevent the subject from being able to cooperate with testing.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Feasibility to selectively stimulate and record from A-delta nerve fibers using the intra-epidermal stimulation electrode as measured by electromyography (EMG) | one year
  Stimulate and record from A-delta nerve fibers in normal individual using intra-epidermal stimulation electrode.

CONTACTS AND LOCATIONS:
Overall Officials: David Walk, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States